CLINICAL TRIAL: NCT03404037
Title: Serum Endostatin Level as a Marker for Coronary Artery Calcification in Type 2 Diabetic Patients With Coronary Heart Disease
Brief Title: Serum Endostatin Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Hazem Mohamed Elashmawy, Professor of Internal Medicine, Zagazig University
Other Study IDs: 3527/20-2-2017
Record Dates: First submitted 2018-01-11; First posted 2018-01-19 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2018-01

CONDITIONS: Diabetes Mellitus, Type 2; Coronary Artery Disease; Coronary Arteriosclerosis
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: Fifty-five coronary artery disease patients without type 2 DM
  Interventions: Diagnostic Test: serum endostatin level
- Group II: Fifty-five coronary artery disease patients with type 2 DM
  Interventions: Diagnostic Test: serum endostatin level

INTERVENTIONS:
Diagnostic Test: serum endostatin level — An oral (metoprolol 20 mg) was given to the patients with heart rates > 60 beats/minute and had no contraindications to beta-blockers, one hour before the scan. Sublingual nitroglycerin was given to all patients before CT examination. A 64-slice CT scanner (Sensation 64; Siemens Medical System, Germany) was used for imaging all subjects. All CT examinations were done during inspiratory breath holding.
  Endostatin levels were measured using a sandwich ELISA kit according to the manufacturer's instructions endostatin ELISA kit (R&D Systems, Minneapolis, Minnesota, USA
  Other Names: Computed tomography

SUMMARY:
To assess the relationship between serum endostatin (ES) and Coronary artery calcification (CAC) in type 2 diabetic (T2DM) patients.

DETAILED DESCRIPTION:
elevated serum endostatin levels were independently associated with increased risk, severity and progression of coronary artery calcification independent of traditional cardiovascular disease risk factors in T2DM subjects with known coronary artery disease. So, Measurement of serum ES levels can improve the diagnosis of coronary artery calcification and could be useful as a high sensitive marker for the presence and progression of atherosclerosis in T2DM patients.

ELIGIBILITY:
Inclusion Criteria: - Patients were between the ages of 50 and 70 years at enrollment.

* Symptomatic or previously recognized coronary artery disease for all the study population.
* Type 2 diabetic patients with the onset of type 2 diabetes occurred at age 30 years or older with no history of ketoacidosis for group II subjects.

Exclusion Criteria:

* left ventricular ejection fraction (LVEF) ≤40%, chronic heart failure, unstable angina, Myocardial infarction, arrhythmia, valvular heart disease, coronary artery bypass surgery, and history of stent placement, liver diseases, malignancy, glomerular filtration rate index < 35 mL/min/m2, serum creatinine level above 4.5 mg/dL, body mass index >30 kg/m2 or < 15 kg/m2, pulmonary edema, stroke, acute infections, severe trauma, recent surgery, inflammatory conditions, thyrotoxicosis, pregnancy and known allergic reactions.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: One hundred ten out documented CAD subjects were divided into two groups; group I (Fifty-five CAD patients without T2DM) and group II (Fifty-five CAD patients with T2DM) addmitted to Zagazig University hospital. Egypt
Sampling Method: Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2017-03-02 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Serum Endostatin Level as a Marker for Coronary Artery Calcification in Type 2 Diabetic Patients with Coronary Heart Disease | 3-Months
  Measurement of serum endostatin and Coronary artery calcification in type 2 diabetic patients patients and non-diabetic patients.

CONTACTS AND LOCATIONS:
Overall Officials: Hazem M Elashmawy, MD. Msc, Principal Investigator — Faculty of medicine, Zagazig University
Locations (1):
- Zagazig University, Faculty of Medicine, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No